CLINICAL TRIAL: NCT03052842
Title: A Phase 2, Single-blind, Randomized, Placebo-controlled Study to Evaluate the Microbiology, Safety and Tolerability of C16G2 Strip Administered in Multiple Doses to Adolescent and Adult Dental Subjects
Brief Title: A Study to Evaluate the Microbiology, Safety and Tolerability of C16G2 Dental Strip Application
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Armata Pharmaceuticals, Inc. (Industry)
Collaborators: Vantage Data Designs, Inc. (Industry); E Squared Trials and Registries, Inc. (Industry); Agility Clinical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: C3J16-S205-00
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Results first posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Three dose groups will be enrolled in an ascending dose escalation manner
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1A: 9.2 mg C16G2 (Experimental): Study subjects will be randomized to receive 9.2 mg C16G2 Strip or Placebo in a 4:1 allocation ratio (8 C16G2 Strip subjects: 2 Placebo Strip subjects). Study arm will be fully enrolled (i.e., the last subject in an arm has completed Visit 3) before enrollment is initiated in the next study arm.
  Interventions: Drug: C16G2 Strip
- Arm 1B: 9.2 mg Placebo (Placebo Comparator): Study subjects will be randomized to receive 9.2 mg C16G2 Strip or Placebo in a 4:1 allocation ratio (8 C16G2 Strip subjects: 2 Placebo Strip subjects). Study arm will be fully enrolled (i.e., the last subject in an arm has completed Visit 3) before enrollment is initiated in the next study arm.
  Interventions: Other: Placebo Strip
- Arm 2A: 18.4 mg C16G2 (Experimental): Study subjects will be randomized to receive 18.4 mg C16G2 Strip or Placebo in a 4:1 allocation ratio (8 C16G2 Strip subjects: 2 Placebo Strip subjects). Study arm will be fully enrolled (i.e., the last subject in an arm has completed Visit 3) before enrollment is initiated in the next study arm.
  Interventions: Drug: C16G2 Strip
- Arm 2B: 18.4 mg Placebo (Placebo Comparator): Study subjects will be randomized to receive 18.4 mg C16G2 Strip or Placebo in a 4:1 allocation ratio (8 C16G2 Strip subjects: 2 Placebo Strip subjects). Study arm will be fully enrolled (i.e., the last subject in an arm has completed Visit 3) before enrollment is initiated in the next study arm.
  Interventions: Other: Placebo Strip
- Arm 3A: 36.8 mg C16G2 (Experimental): Study subjects will be randomized to receive 36.8 mg C16G2 Strip or Placebo in a 4:1 allocation ratio (8 C16G2 Strip subjects: 2 Placebo Strip subjects).
  Interventions: Drug: C16G2 Strip
- Arm 3B: 36.8 mg Placebo (Placebo Comparator): Study subjects will be randomized to receive 36.8 mg C16G2 Strip or Placebo in a 4:1 allocation ratio (8 C16G2 Strip subjects: 2 Placebo Strip subjects).
  Interventions: Other: Placebo Strip

INTERVENTIONS:
Drug: C16G2 Strip — Antimicrobial Peptide
  Arms: Arm 1A: 9.2 mg C16G2; Arm 2A: 18.4 mg C16G2; Arm 3A: 36.8 mg C16G2
Other: Placebo Strip — Placebo
  Arms: Arm 1B: 9.2 mg Placebo; Arm 2B: 18.4 mg Placebo; Arm 3B: 36.8 mg Placebo

SUMMARY:
Single-blind study to evaluate whether C16G2 Strip administered in multiple doses can effectively kill the bacteria in the oral cavity that cause dental caries..

DETAILED DESCRIPTION:
A single-blind, randomized, placebo-controlled, phase 2 study to evaluate oral microbiology and safety of multiple C16G2 Strip applications in male and female dental subjects 12-75 years of age.

The study will compare multiple study drug administrations of 9.2 mg, 18.4 mg, and 36.8 mg C16G2 Strip or Placebo in Study Arms 1 through 3, respectively. Enrollment of subjects in Study Arms 1 through 3 will occur sequentially in an ascending dose-escalation manner. Before dosing of study drug, eligible subjects will receive professional dental prophylaxis between Days -7 and -2. Subjects will receive 11 doses administered over approximately two weeks. Each subject will receive a single dose on Day 0, followed by 5 days of AM and PM dosing starting on Day 7. To evaluate the durability of S. mutans suppression, study subjects will be followed for microbiology for up to 1 month after the last study drug administration.

Clinic visits include Visit 1 (Screening/Days -30 to -1), Visit 2 (Prophylaxis/Day -7 to -2), Eligibility Confirmation & Baseline Visit 3, Follow-up Visits 4-7 (Safety and Microbiology), Visits 8-17 (Study Drug Administration), Follow-up Visits 18-20 (Safety and Microbiology) and Follow-up Visits 21-22 (Microbiology only).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 12-75 years of age
2. Adults subjects provide written informed consent and adolescent subjects give written or verbal assent, as appropriate, and parent(s) or legal guardian(s) give written informed consent
3. Female subjects of childbearing potential must agree to use one of the following forms of contraception from screening through the last study visit: hormonal (oral, implant, or injection) begun >30 days prior to screening; barrier (condom, diaphragm, or cervical cap with spermicide); intrauterine device (IUD). Acceptable contraceptive options may also include abstinence, relationship with a same sex partner or partner who has had a vasectomy at least six (6) months prior to the screening visit
4. Negative urine pregnancy test in all females of childbearing potential (past menarche)
5. Male subjects of sexual activity age: willing to use contraception or abstain from sexual activity beginning with the first exposure to study drug and continuing until discharged from the study due to completion or Early Termination
6. Healthy, as determined by the Investigator (in consultation with the Medical Monitor, as needed), based on medical and dental history, concurrent illnesses, laboratory results, concomitant medications, oral cavity assessment, and targeted physical examination (general, extraoral, head and neck) during Screening Note: Subjects on a stable dose of medication may be eligible for screening and will be assessed by the medical monitor on a case-by-case basis.
7. Have a minimum of 12 bicuspids and molars with a minimum of 8 molars and bicuspids NOT having restorations, crowns or sealants
8. Demonstrated ability to expectorate ≥2 mL of stimulated saliva in 5 minutes
9. Have a salivary S. mutans of 1.0 x 10^5 CFUs/mL or greater at Screening using mitis salivarius-bacitracin (MSB) agar plating
10. Willing to refrain from using non-study dentifrice and other non-study oral care products (oral care rinses, fluoride products, etc.) during the study
11. Willing to postpone elective dental procedures (e.g., dental cleanings) between Screening and final post-treatment visit (End of Study or Early Termination)
12. Willing and able to comply with oral hygiene and diet instructions
13. Able to communicate with the Investigator/study center personnel, understand and comply with the study requirements, and willing to return for protocol-specified visits at the appointed times

Exclusion Criteria:

1. Advanced periodontal disease
2. Active caries lesion(s) within 30 days prior to study drug administration (confirmed by comprehensive caries examination including standard radiographs). Subjects presenting with insipient, non-cavitated lesion(s) are not excluded Note: If radiographs are deemed appropriate for the study and taken within 6 months prior to the Screening visit, these may be used for determining eligibility and are not required to be repeated at Screening
3. Partially erupted teeth where the entire crown is not erupted or an operculum is present
4. Medical condition (e.g., artificial heart valve, history of infective endocarditis, cardiac transplant with valvular dysfunction, congenital heart disease or total joint replacement) for which antibiotics are recommended prior to dental visits and/or procedures
5. Pathologic lesions of the oral cavity (suspicious or confirmed)
6. Full dentures or permanent orthodontic appliances, e.g., braces, buccal or lingual brackets.
7. Use of systemic antibiotics, topical oral antibiotics, or use of other drugs, which in the opinion of the Investigator could influence the study outcome, beginning 30 days prior to Screening until the end of study participation
8. Medical history indicating the woman is pregnant, breastfeeding/lactating or has a positive urine pregnancy test
9. Participation in a clinical trial or receipt of a non-FDA approved therapy within 30 days prior to study drug administration (depending on the specifics, participation in an observational study is not necessarily excluded)
10. Presence of any condition or concurrent illness, which in the opinion of the Investigator, would compromise normal immune function (e.g., diabetes, rheumatoid arthritis, lupus, liver disease, organ transplant, etc.), interfere with the use of study dentifrice and oral care products, or interfere with the ability to comply with study requirements, or jeopardize the safety of the subject or the validity of the study results

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pittaway, DMD, Principal Investigator — Plaza West II Dental Group
Locations (3):
- United States (3):
  - John F. Pittaway, DMD, Kalispell, Montana
  - Jacqueline Kleven, DDS, Bedford, Texas
  - Anthony Henegar, DDS, PA, Irving, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Group: Pooled Placebo: Subjects enrolled in Arms 1B (N=2), 2B (N=2) and 3B (N=2) were pooled into one group.
Period: Overall Study
Arm/Group | Arm 1A: 9.2 mg C16G2 | Arm 2A: 18.4 mg C16G2 | Arm 3A: 36.8 mg C16G2 | Group: Pooled Placebo
Started | 8 | 8 | 8 | 6
Completed | 8 | 8 | 8 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 2A: 18.4 mg C16G2: Study subjects will be randomized to receive 18.4 mg C16G2 Strip or Placebo in a 4:1 allocation ratio (8 C16G2 Strip subjects: 2 Placebo Strip subjects). Study arm will be fully enrolled (i.e., the last subject in an arm has completed Visit 3) before enrollment is initiated in the next study arm.
  Placebo Strip: Placebo
- Total: Total of all reporting groups
Arm/Group | Arm 1A: 9.2 mg C16G2 | Arm 2A: 18.4 mg C16G2 | Arm 3A: 36.8 mg C16G2 | Group: Pooled Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 30
Age, Continuous [Mean (Full Range); unit: years] — Population: N=8: Participants who received 9.2mg C16G2, 18.4mg C16G2, and 36.8mg C16G2, respectively N=6: placebo particpants from 3 arms
  years | 26.2 [18 to 54] | 26.2 [18 to 41] | 31.1 [17 to 55] | 23 [17 to 55] | 26.9 [14 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 4 | 3 | 16
  Male | 3 | 4 | 4 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 1 | 1 | 7
  Not Hispanic or Latino | 7 | 4 | 7 | 5 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Antimicrobial Activity of C16G2
Description: To assess the targeted antimicrobial activity of C16G2 applications as measured by a reduction in Streptococcus mutans in saliva and dental plaque using S. mutans CFUs using mitis-salivarius bacitrain (MSB) agar plating. Streptococcus species present in the oral cavity have been traditionally isolated from oral cavity samples using MSB agar plates. The antimicrobial activity of crystal violet dye, high sucrose content, sodium tellurite and bacitracin effectively prevent the growth of all bacteria except for streptococci. Further differentiation of streptococci is accomplished by observing colony morphology. S. mutans grows in large blue colonies with dry frosted tops or pale blue gumdrops and can be differentiated from other bacterial colonies.
Time Frame: Measured up to 1 months post last study drug administration
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Arm 1A: 9.2 mg C16G2 | Arm 2A: 18.4 mg C16G2 | Arm 3A: 36.8 mg C16G2 | Group: Pooled Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6
CFU/mL
  Saliva Sample: S. mutans Change from Baseline to Visit 22 | -0.2 (1.16) | -0.04 (0.79) | 0.005 (0.34) | 0.15 (0.41)
  Dental Plaque Sample: S. mutans Change from Baseline to Visit 22 | 0.14 (0.93) | -0.19 (1.09) | 0.36 (0.29) | 0.24 (1.02)

2. Primary Outcome: Total Oral Bacterial Levels
Description: To assess total bacteria in saliva and dental plaque post study drug administration using total bacteria CFUs using Todd Hewitt (TH) agar plating and the log transformed changes from baseline Total Bacteria levels in dental plaque and saliva including N, mean, SD, median and range at each assessment time point following the first administration of C16G2.
Time Frame: Measured up to 1 months post last study drug administration
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Arm 1A: 9.2 mg C16G2 | Arm 2A: 18.4 mg C16G2 | Arm 3A: 36.8 mg C16G2 | Group: Pooled Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6
CFU/mL
  Saliva Sample - Total Bacteria by TH Agar Plating from Baseline to Visit 22 | 0.28 (0.38) | 0.33 (0.40) | 0.26 (0.22) | 0.30 (0.64)
  Dental Plaque Sample - Total Bacteria by TH Agar Plating from Baseline to Visit 22 | 0.46 (0.49) | 0.10 (0.89) | 0.53 (0.42) | 0.08 (0.94)

3. Secondary Outcome: To Evaluate the Safety and Tolerability of Multiple C16G2
Description: Safety will be assessed by performing targeted physical examinations, oral cavity exams, taking vital signs and collection of adverse events categorized according to system organ class (SOC) and preferred term (PT) based on coding to the Medical Dictionary for Regulatory Activities (MedDRA®), Version 17.1. Comprehensive examinations of oral hard and soft tissue structures, as well as targeted exams of specific musculoskeletal and extraoral sites were performed at selected time points; vital signs (blood pressure, heart rate and temperature) were taken.
Time Frame: Up to 1 week post last study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A: 9.2 mg C16G2 | Arm 2A: 18.4 mg C16G2 | Arm 3A: 36.8 mg C16G2 | Group: Pooled Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6
Participants
  Participants with Adverse Events Related to Study Drug | 0 | 0 | 0 | 0
  Participants with Clinical Significant Oral Cavity Changes | 0 | 0 | 0 | 0
  Participants with Clinical Significant Vital Sign Changes | 0 | 0 | 0 | 0
  Participants with Abnormal Physical Exam Findings | 0 | 0 | 0 | 0
  Participants with Completed Study | 8 | 8 | 8 | 6

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Arm 1A: 9.2 mg C16G2 | Arm 2A: 18.4 mg C16G2 | Arm 3A: 36.8 mg C16G2 | Group: Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT03052842/Prot_SAP_000.pdf